CLINICAL TRIAL: NCT04335981
Title: A Randomized, Single-Center Study to Determine Swallow Outcomes in Subjects With Head and Neck Lymphedema Receiving Early Intervention With Pneumatic Compression
Brief Title: Determining Swallow Outcomes in Head & Neck Lymphedema Subjects Receiving Early Intervention With Pneumatic Compression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than anticipated enrollment.
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 8020
Record Dates: First submitted 2020-03-10; First posted 2020-04-07 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Head and Neck Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FT-CC and Swallow Exercises (Experimental)
  Interventions: Device: FT-CC and Swallow Exercises
- Swallow Exercises (Active Comparator)
  Interventions: Other: Swallow Exercises

INTERVENTIONS:
Device: FT-CC and Swallow Exercises — Once daily treatment with FT Plus with investigational connectivity software and standard of care swallow exercises.
  Arms: FT-CC and Swallow Exercises
Other: Swallow Exercises — Standard of care swallow exercises.
  Arms: Swallow Exercises

SUMMARY:
The objective of the study is to assess the effect early pneumatic compression (prior to confirming cancer-free status via PET or CT imaging) has on swallow outcomes, positron emission tomography (PET) measurements, function, and complication rate post-radiotherapy in subjects treated for oropharyngeal cancer.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, two-arm, wait-list control study that plans to enroll a total of 24 subjects in the United States. A baseline screening will take place where all subjects who provide consent and meet the eligibility criteria following completion of radiotherapy will begin a 6 weeks regimen of in-home swallow exercises. They will then return to the clinic for final screening and randomization into one of two treatment groups: Flexitouch Plus Cellular Connectivity (FT-CC) and Swallow Exercises (Intervention) or Swallow Exercises alone (Standard Care). A total of 3 in-clinic visits and 1 phone call will be conducted over a 12-week period. The Standard Care group will be offered an optional 6 week follow-up period to use the device in-home and will be seen in the clinic for one additional follow-up Visit 2. A reading center with personnel blinded to treatment assignment will be used to interpret the MBS and PET study results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. A previous diagnosis of oropharyngeal carcinoma requiring treatment with radiation therapy
3. Diagnosis/evidence of lymphedema stage 1a or higher by clinical presentation based upon MD Anderson Cancer Center Head and Neck Lymphedema rating scale
4. EAT-10 score >4 at Baseline and Randomization Visits (prior to randomizing subject)
5. The head and neck garments must fit appropriately (for patients with a tracheostomy, the fit will be assessed to ensure that the garments do not interfere with their tracheostomy)
6. Ability to perform swallow exercises
7. Willing and able to comply with the study protocol requirements and all study-related visit requirements
8. Willing and able to provide informed consent prior to study participation

Exclusion Criteria:

1. Synchronous treatment for cancer (may or may not have successfully complete prior cancer treatment)
2. Other known causes of dysphagia such as previous radiation to the head and neck, or neuromuscular or neurodegenerative known to have a strong association with dysphagia (i.e., Parkinsons, ALS, MS, OPMD)
3. Poorly controlled: kidney disease (glomerular filtration rate < 30 mls per minute), hypoproteinemia, pulmonary hypertension, hypothyroidism or parathyroidism, cyclic edema, or Munchausen Syndrome (for which endocrinologist recommends against neck compression)
4. Carotid sinus hypersensitivity syndrome
5. Symptomatic carotid artery disease, as manifested by a recent transient ischemic attack (within 30 days), ischemic stroke, or amaurosis fugax (monocular visual ischemic symptoms or blindness)
6. Symptomatic bradycardia in the absence of a pacemaker
7. Internal jugular venous thrombosis (within 3 months)
8. Increased intracranial pressure or other contraindications to internal or external jugular venous compression
9. Acute radiation dermatitis, unhealed surgical scar, unhealed or open wounds, surgical flap less than 6-8 weeks post-operative
10. Facial or head and neck dermal metastasis
11. Acute infection/inflammatory disease of the head and neck region (e.g., facial infection, parotid gland abscess, acute cellulitis, or other uncontrolled skin/untreated head and neck inflammatory skin disease)
12. Any condition in which increased venous and lymphatic return is undesirable
13. Heart failure (acute pulmonary edema, decompensated acute heart failure)
14. Subject is pregnant or trying to become pregnant
15. Acute venous disease (acute thrombophlebitis, acute deep venous thrombosis, acute pulmonary embolism)
16. The subject has comorbidities which, in the opinion of the investigator, will not be appropriate for the study or the subject has an estimated life expectancy of less than 1½ months
17. Any subject who is considered to be part of a vulnerable population (e.g., prisoners or those without sufficient mental capacity)
18. The subject has participated in any investigational drug or device research study within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Swallow outcomes via modified barium swallow - Penetration-Aspiration Scale (PAS) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  PAS is an eight-point ordinal severity scale scoring the depth of airway invasion by the bolus, whether it is expelled from the airway as well as any patient reaction. It ranges from one (material does not enter the airway) to eight (material enters the airway, passes below the vocal folds, and no effort is made to eject). Min value = 1, Max value = 8, the lower the score the better.
Swallow outcomes via modified barium swallow - Pharyngeal Constriction Ratio (PCR) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  PCR is calculated by dividing the pharyngeal area (cm2) of the bolus hold frame (PAHOLD) by the maximum pharyngeal contraction frames (PAMAX). Min value = 0, Max value = 1. The lower the score, the better the outcome.
Swallow outcomes via modified barium swallow - Upper Esophageal Sphincter Opening (UESmax) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  UES measurements will include the: (1) maximum width of the UES opening as defined by the line between the anterior and posterior walls of the pharyngoesophageal segment at its narrowest area during its maximum opening in a lateral view, and (2) the maximum width of the UES opening as viewed anteriorly. Min value = 0, max value = 2. Greater the score, the better the outcome.
Swallow outcomes via modified barium swallow - Esophageal Bolus Transit Time (ETT) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  The time it takes the bolus to get through the cricopharyngeal muscle (where the esophageal phase is initiated) to the bottom of the esophagus (at the junction of the lower esophageal sphincter). Min value = 0, max value = 60. The lower the score, the better the outcome (seconds).
Swallow outcomes via modified barium swallow - Normalized residue ratio scale (NRRS) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Pharyngeal residue is the term used to describe material that remains in the pharynx post swallow (also called retention or stasis). The NRRS is calculated using ImageJ pixel area measures of residue in the valleculae. Min value = 0, max value = 1. The lower the score, the better the outcomes.
Swallow outcomes via modified barium swallow - Posterior Pharyngeal Wall Thickness (PPW) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  PPW is the thickness of the posterior pharyngeal wall in lateral view while holding a 1-ml liquid bolus in oral cavity prior to swallow (PPWhold). Min value = 0, max value = 30. The lower the score the better the outcomes (mm)
Function - Stimulated Saliva Secretion Rate | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Stimulated Saliva Secretion Rate is the measure of total saliva collected in 3 minutes while chewing gum.
Swallow outcomes via patient reported outcome measure - Eating Assessment Tool (EAT-10) Questionnaire Score | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Min value = 0, max value = 4. The lower the score the better the outcome.
Patient Reported Function - Voice Handicap Index (VHI-10) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  A survey that quantifies the functional, physical, and emotional impacts of a voice disorder on a subject's quality of life. It captures the subject's subjective rating of a series of 10 questions. Min value = 0, max value = 40. The lower the score the better the outcomes.
Patient Reported Function - Functional Assessment of Cancer Therapy - Head and Neck (FACT HN) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  A survey which inquires on a series of concerns related to the head and neck region including oral comfort, breathing, voice, eating, appearance, tobacco, alcohol, and communication. The subject is asked to indicate how important each of the 39 listed concerns have been in the past 7 days. Min value = 0, max value = 148. The higher the score the better the quality of life.
Nutrition - Weight | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Weight
Nutrition - Body Mass Index (BMI) | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  BMI
Complications - Treatment Interruptions | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Number/days of treatment interruptions
Complications - Hospitalizations | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Number/days of hospitalizations
Complications - Pulmonary Infections | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Number/days of pulmonary infections
Complications - Adverse Events | Changes between Baseline, 6-Week Follow-Up, 12-Week Follow-Up, and 18-Week Follow-Up
  Total number of adverse events

OTHER OUTCOMES:
PET Measurements - Epiglottic Thickness | Changes between Baseline and 12-Week Follow-Up
  A measurement of the epiglottic thickness.
PET Measurements - Prevertebral Space | Changes between Baseline and 12-Week Follow-Up
  A measurement of the prevertebral space.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California - Davis, Sacramento, California, United States